CLINICAL TRIAL: NCT03940365
Title: Fetal Life: Calibration, Noninferiority and Feasibility Studies for Smart-Device Based Uterine Activity Monitoring
Brief Title: Fetal Life: Smart-Device Based Uterine Activity Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fetal Life LLC (Industry)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19.0011
Record Dates: First submitted 2019-04-11; First posted 2019-05-07 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Labor Pain; Contraction
Keywords: Labor; Uterine contraction
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The study will use a single group for the intervention as detailed above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): As detailed above, a single group will be used for the study to compare the output of the study device with the output of the standard device in each patient.
  Interventions: Device: Fetal Life tocometer device

INTERVENTIONS:
Device: Fetal Life tocometer device — The fetal life tocometer device is a uterine contraction monitor which is less expensive to manufacture than existing contraction monitor devices and which pairs with a smart device rather than a bulky output device.

SUMMARY:
This study will compare the performance of a contraction monitor (tocometer) device developed by Fetal Life with standard tocometer devices.

The study aims to test a uterine contraction monitor that can be applied by the patient to her abdomen and connected to her smart device to detect the frequency and duration of uterine contractions. Phase 1 will collect data for calibration of the monitor and for a noninferiority study comparing the Fetal Life uterine contraction monitor (tocometer) with standard tocometry devices. Phase 2 will be a feasibility study in which patients will position the monitor, connect to the corresponding Fetal Life app and measure their own uterine contraction activity.

The study's hypothesis is that after calibration, the new monitor will reliably detect at least 95% of the number and duration of contractions detected by the standard monitor, and that the device will perform comparably whether applied by the patient or by research staff.

DETAILED DESCRIPTION:
Pregnant patients are counseled to monitor the frequency and duration of contractions in order to know when to come to the hospital for evaluation. Once a pregnant patient arrives at the hospital, contraction monitoring is important to help diagnose labor, which is defined as contractions with cervical change. In the hospital, a pressure-sensitive external contraction monitor or tocometer is positioned on the patient's abdomen with a belt to measure the frequency and length of her contractions. These tocometry monitors are impractical for home use because of their expense and because they create their output by connecting to bulky component devices. For these reasons reason, pregnant patients at home do not have access to automated tocometry monitoring.

Patients are educated during prenatal care that contractions should be timed from the start of one contraction to the start of the next. These instructions can be difficult for patients to remember, and patients who are having painful contractions may prefer a more automated method for timing contractions. All methods currently available for home contraction tracking (on paper, using a smart device, or using one of many available smart device applications) require manual data entry either by the patient or her support partners.

Patients are cautioned during pregnancy to maintain awareness of the development of uterine contractions. Early in pregnancy, patients are frequently counseled that infrequent, irregular contractions can be normal, but that frequent contractions occurring in a pattern can be a sign of preterm labor. As dehydration can cause the uterus to contract, preterm patients who notice contractions occurring in a pattern are often instructed to drink water, observe their contraction pattern, and come to the hospital if their contractions continue to occur every 15 minutes or more frequently following oral hydration. At term, patients are frequently counseled to come to the hospital when they are experiencing contractions that last about a minute, are occurring every five minutes, and have been at this duration and frequency for about an hour. Both preterm and at term, patients may have runs of contractions which resolve with time and hydration, but patients in both situations need to recognize when their contractions have reached the parameters recommended by their health care providers to seek medical attention.

The new tocometer device tested in this study has significant cost savings in comparison to existing devices, and connects to a smart phone or tablet rather than a bulky receiver. The device will allow the patient to apply a monitor belt, connect it to her smart phone, and view a graphical representation of her contraction pattern with verbal descriptors that she can share with her health care team. Many patients have at least one visit to the hospital for evaluation of a contraction pattern which did not warrant this time and expense. This device may help patients to share a more accurate report of their symptoms with their prenatal care providers, potentially decreasing the stress of manual contraction tracking, improving the understanding of progress in early labor and decreasing unnecessary hospital visits. The device and app will not give the patient instructions on whether to come to the hospital, but will be used to help the patient understand if her uterine activity meets the parameters her prenatal care provider has given her to come in for evaluation. The Fetal Life device is constructed of smooth, latex-free plastic, is powered by a Lithium battery similar to a watch battery, and is held in place using a standard tocometry belt manufactured by General Electric. The investigators consider this to be a nonsignificant risk device.

Phase 1 of this initial trial will allow a noninferiority comparison of the performance of this new contraction monitoring device with standard devices currently used in Labor and Delivery settings for monitoring duration and frequency of contractions. Phase 2 will assess feasibility for patient use.

Procedure for Calibration and Noninferiority Phase (Phase 1):

* Patients meeting inclusion criteria will be offered participation in the study by the Clinical Trials Unit (CTU) Staff
* If the patient agrees to participate, CTU staff will obtain consent.
* The patient will be assigned a participant number.
* The Fetal Life tocometer will be applied to the patient's lower abdomen in addition to the standard tocometer used on Labor and Delivery and secured with the monitor belt by CTU staff
* The Fetal Life tocometer will be paired the study iPad and output will be captured by CTU staff
* The patient will be asked to cough in order to create a peak that synchronizes the graphic output of the Fetal Life tocometer and the standard tocometer
* The patient will be monitored with the both the standard tocometer and the Fetal Life tocometer for 45-60 minutes
* If the maternal or fetal status requires changes of maternal position during the trial, the Fetal Life monitor may be left in place, disconnected from the iPad or removed from the patient, whichever is least disruptive, so as not to interfere with the patient's obstetrical care in any way
* CTU staff will document patient's age, parity, estimated gestational age and body mass index on a data collection sheet identified by participant number. No personal health information will be maintained on the data sheet.
* If 45-60 minutes of monitoring is not completed, CTU staff will document the reason why
* Patient will complete a brief survey on monitor comfort in comparison to the standard monitor
* Image files from the standard tocometry fetal monitoring system will be exported for comparison with the output of the Fetal Life tocometer.
* Fetal Life device will be sanitized with the antiviral, antibacterial wipes used routinely for sanitation of the standard tocometer devices before use with another patient. A new belt will be attached to the device for each subject.
* For calibration, deidentified data from standard tocometer and the Fetal Life device will be reviewed by the team in the University of Louisville School of Engineering so that any needed adjustments can be made to the pressure transducer's sensitivity or graphic output
* After calibration is completed (estimate 3 subjects needed), subjects will then be enrolled using the same protocol to collect data required for statistical analysis of non-inferiority

Procedure for Feasibility Phase (Phase 2):

* Patients meeting the inclusion criteria will be offered participation in the study by the Clinical Trials Unit (CTU) Staff
* If the patient agrees to participate, CTU staff will obtain consent.
* The patient will be assigned a participant number.
* The patient will read the Fetal Life monitor instructions
* Standard tocometry and fetal heart rate devices will be removed
* The patient will apply the Fetal Life monitor using the positioning belt and will connect to the study iPad or lap top computer via Bluetooth
* Fifteen minutes of monitoring will be captured via the iPad or lap top computer by CTU staff
* During this time, the patient will note when she perceives the beginning and the end of her contractions; this will be documented the Clinical Trials Unit staff with time notations
* Fetal Life monitor will be removed and the standard external fetal monitoring will resume
* Patient will complete the patient survey

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients on the Labor and Delivery unit
* Contracting every five minutes or more frequently by standard tocometry monitor
* Category 1 fetal heart tracing (reassuring tracing with moderate variability and no decelerations)
* Cervical examination completed and awaiting repeat examination in 2-4 hours
* 37 weeks or greater
* Singleton pregnancy (not multiple gestation)
* Live fetus
* Undergoing tocometry monitoring with standard devices
* English speaking
* Age between 20 years and 40 years

Exclusion Criteria:

* Nonreassuring fetal heart tracing
* Any active skin lesions or infections

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of contractions measured by Fetal Life tocometer in comparison with standard tocometer | one hour of monitoring per subject
  number of contractions and duration in seconds
Duration of contractions measured by Fetal Life tocometer in comparison with standard tocometer | one hour of monitoring per subject
  number of contractions and duration in seconds
Physical comfort of device in comparison with standard monitor | Survey on completion of one hour of monitoring
  Patient survey question: is the study device (black rectangle) more comfortable, less comfortable of the same in comfort as the routine monitor (white disk)?
Stability of device placement on abdomen in comparison with standard monitor | Survey on completion of one hour of monitoring
  Patient survey question: does the study device (black rectangle) stay where it positioned on your abdomen when you move around better than the routine monitor (white disk), less that the routine monitor or about the same as the routine monitor?
Preference for device over standard monitor | Survey on completion of one hour of monitoring
  Patient survey question: do you any preference for study device (black rectangle), the routine monitor (white disk) or no preference between the two?
Were directions clear to patient? | Survey completed by subject on completion of 15 minutes of monitoring
  Patient survey question: did you understand the direction for using the device? (yes/no)
Was patient able to position the device? | Survey completed by subject on completion of 15 minutes of monitoring
  Patient survey question: were you able to position the device on your abdomen? (yes/no)
Was patient able to pair the device with the app? | Survey completed by subject on completion of 15 minutes of monitoring
  Patient survey question: were you able to pair the device with the smart device app? (yes/no)
Was patient able to see their contractions on the app? | Survey completed by subject on completion of 15 minutes of monitoring
  Patient survey question: were you able to see your contractions on the smart device app? (yes/no)
Did contractions on the app correlate with the patient's experience? | Survey completed by subject on completion of 15 minutes of monitoring
  Patient survey question: did the information visible on the smart device app accurately reflect the contractions you were feeling? (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Petruska, MD, Principal Investigator — University of Louisville
Locations (1):
- University Hospital, University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis D, Downe S; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Intermittent auscultation. Int J Gynaecol Obstet. 2015 Oct;131(1):9-12. doi: 10.1016/j.ijgo.2015.06.019. No abstract available. PMID 26433400
- [Background] Hoffman E.B., Sen, P.K., Weinberg, C.R. Within-cluster resampling. Biometrika (2001), 88(4): 1121-1134.
- [Background] Lorenz DJ, Levy S, Datta S. Inferring marginal association with paired and unpaired clustered data. Stat Methods Med Res. 2018 Jun;27(6):1806-1817. doi: 10.1177/0962280216669184. Epub 2016 Sep 20. PMID 27655806